CLINICAL TRIAL: NCT02104856
Title: Bronchial Thermoplasty (BT) Global Registry
Brief Title: Bronchial Thermoplasty Global Registry
Acronym: BTGR
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: E7086
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Asthma
Keywords: Asthma; Bronchial Thermoplasty; Registry; Device; Alair
MeSH Terms: conditions — Asthma | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Alair System (Bronchial Thermoplasty): Asthma patients undergoing Bronchial Thermoplasty treatment with commercially available Alair device as per Directions For Use.
  Interventions: Device: Alair System (Bronchial Thermoplasty)

INTERVENTIONS:
Device: Alair System (Bronchial Thermoplasty)

SUMMARY:
The primary objective of this Registry is to collect real-world data on patients undergoing bronchial thermoplasty (BT) treatment.

DETAILED DESCRIPTION:
This Registry is a prospective, open-label, single arm, observational registry to collect outcome data as well as clinical and demographic characteristics of patients undergoing BT treatment in the "real world" setting. Patients will be recruited at participating study centers that offer BT as a treatment option to patients with asthma who remain symptomatic despite taking standard of care maintenance medications.

The Registry will be conducted at up to 80 sites globally and will enroll up to 500 patients. The treatment period is from the date of the first BT procedure until 6 weeks after the third (last) procedure (approximately 12 weeks). The post-treatment period starts at the date of the 6-week follow up visit after completion of the third (last) BT procedure for 2-years of follow-up.

The primary endpoint will be the proportion of patients who experience severe asthma exacerbations at 1 and 2 years following BT treatment with the Alair System.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an adult aged 18 years or older and is scheduled to undergo BT treatment according to the Alair System DFU.
2. Patient is able to read, understand, and sign a written Informed Consent to participate in the Registry and able to comply with the registry requirements.

Exclusion Criteria:

1. Patient has any medical condition that would make them inappropriate for BT treatment, in the Investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing BT according to labeled indications will be approached to participate in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience severe asthma exacerbations | 2 years
  The primary endpoint will be the proportion of patients who experience severe asthma exacerbations at 1 and 2 years following BT treatment with the Alair System.

SECONDARY OUTCOMES:
Asthma Quality of Life Questionnaire (AQLQ) score | 2 years
  Change from baseline in Asthma Quality of Life Questionnaire (AQLQ) scores will be summarized descriptively for Year 1 and Year 2 post-BT.
Asthma Control Test (ACT) score | 2 years
  Change from baseline in Asthma Control Test (ACT) scores will be summarized descriptively for Year 1 and Year 2 post-BT.
Emergency department visits for asthma symptoms | 2 years
  Will be summarized both by the incidence (percentage of subjects reporting at least one event) and event rates (events/subject/year) for 1 and 2 Years post-BT.
Hospitalizations for asthma symptoms | 2 years
  Will be summarized both by the incidence (percentage of subjects reporting at least one event) and event rates (events/subject/year) for 1 and 2 Years post-BT.
Unscheduled office visits including urgent care visits for asthma symptoms. | 2 years
  Will be summarized both by the incidence (percentage of subjects reporting at least one event) and event rates (events/subject/year) for 1 and 2 Years post-BT.
Pre- and post-bronchodilator Forced Expiratory Volume in one minute (FEV1) | 2 years
  Pre- and post-bronchodilator FEV1 will be summarized for Year 1 and Year 2 post-BT treatment (% predicted and absolute value). Change from baseline will also be summarized.
Respiratory Adverse Events | 2 years
  Separated by treatment period and post-treatment period
Lung Volumes | 2 years
  Collected at sites where it is standard of care
Diffusion Capacity | 2 years
  Collected at sites where it is standard of care
Asthma maintenance medication use (Long Acting Beta Agonists, steroids etc.) | 2 years
  Collect asthma maintenance medications at all sites
Patient satisfaction survey score | 2 years
  Two question survey collected at 12 month and 24 month annual visit
Allergic skin test or Radioallergosorbent Test (RAST) (perennial, seasonal, mold) | 2 years
  Collected at sites where it is standard of care
Sputum eosinophils | 2 years
  Collected at sites where it is standard of care
Exhaled nitric oxide (eNO) | 2 years
  Collected at sites where it is standard of care
Methacholine challenge (Methacholine PC20) | 2 years
  Collected at sites where it is standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Robert Niven, MD, Principal Investigator — Wythenshawe Hospital - University of Manchester; Alfons Torrego, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Felix Herth, MD, Principal Investigator — Thoraxklinik University of Heidelberg
Locations (19):
- Australia (3):
  - Macquarie University Private Hospital, North Ryde, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Peninsula Health, Frankston, Victoria
- Klinika Tuberkulozy a Respiracnich Onemocneni, Prague, Czechia
- Germany (4):
  - Universitätsklinikum Bonn, Bonn
  - Ruhrlandklinik, Westdeutsches Lungenzentrum, Essen
  - Thoraxklinik, University of Heidelberg, Heidelberg
  - University Hospital of Regensburg, Regensburg
- Italy (3):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Ancona
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Aricispedale Santa Maria Nuova, Reggio Emilia
- Academic Medical Center, Amsterdam, Netherlands
- University of Cape Town Groote Shuur Hospital, Cape Town, South Africa
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Germans Trias I Puyol, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
- United Kingdom (2):
  - Gartnavel General Hospital, Glasgow, Scotland
  - Wythenshawe Hospital University of Manchester, Manchester

REFERENCES:
- [Derived] Torrego A, Herth FJ, Munoz-Fernandez AM, Puente L, Facciolongo N, Bicknell S, Novali M, Gasparini S, Bonifazi M, Dheda K, Andreo F, Votruba P, Langton D, Flandes J, Fielding D, Bonta PI, Skowasch D, Schulz C, Darwiche K, McMullen E, Grubb GM, Niven R. Bronchial Thermoplasty Global Registry (BTGR): 2-year results. BMJ Open. 2021 Dec 16;11(12):e053854. doi: 10.1136/bmjopen-2021-053854. PMID 34916324